CLINICAL TRIAL: NCT01710618
Title: SEXI: Sciatic Expression and Identification of Differential Proteins in Traumatized Versus Non-traumatized Nerves
Brief Title: SEXI: Sciatic Expression and Identification of Differential Proteins in Traumatized Versus Nontraumatized Nerves
Acronym: SEXI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 359367-12
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Pain
Keywords: Protein Expression of Sciatic Nerve; traumatized sciatic nerve
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sciatic nerve specimen will be obtained
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to elucidate the different proteins that may appear on the "injured" end of the sciatic nerve and compare it to the other end of the cut nerve, which is "uninjured". By comparing the "normal" versus "traumatized" ends of the cut sciatic nerve, the investigators hope to identify proteins that may be specifically related to pain. For instance, if the non-traumatized end of the nerve has none of Protein X but the traumatized end of the nerve has a lot of Protein X, then Protein X would be a protein that the investigators will want to study further and see if it plays any role in the sensation of pain.

Other studies have shown that there are specific pain-related proteins and they may be increased or decreased after traumatic injury. If the investigators are able to identify specific proteins that are related to pain, then that may eventually lead to the development of medications that will block those proteins and decrease the sensation of pain.

DETAILED DESCRIPTION:
Subjects scheduled for final amputation revision and closure(s) will be approached to participate in the study. On the day of the study participant's planned amputation revision, research staff will liaise with surgical staff to coordinate nerve specimen retrieval. If a patient is to have an above the knee amputation, a sciatic nerve specimen will be obtained, if a patient is to have a below the knee or through knee amputation, a tibial nerve specimen will be obtained (the major component of the sciatic nerve after it divides into the tibial and peroneal nerves in the popliteal fossa of the knee). The surgeon will place a suture in the proximal end of the specimen to indicate the non-traumatized end of the nerve, as well as provide an estimate of the longitudinal location of the nerve sampled (i.e. 10cm distal to the knee joint line, 15 cm proximal to the knee at the knee joint level). Each sample will be excised in the same manner - using a scalpel. Once the tissue is excised by the surgeon, it will be placed in a plastic test tube that is labeled with the subjects' study identification number (with the suffix "A" or "B" if two samples are being retrieved from that subject), transferred to a member of the research staff and immediately frozen in liquid nitrogen. The frozen specimen will then be delivered to the Department of Research Programs laboratory where it will be stored at -80°C prior to analysis. The promixal, middle, and distal samples will be obtained at the DRP lab and the remaining segments of nerve will be replaced in the -80 freezer for future analysis. Samples will then be sent to Duke University for processing and analysis via a secure air mail carrier. The task of processing samples will be performed immediately prior to mass spectroscopy analysis by colleagues at Duke University. Collaborator Dr Moseley's lab responsibilities include both protein extraction and assay. The number of extractions per sample will vary depending on its length, from 2 to about 50. Collaborator Dr Van de ven's lab responsibilities include sample handling, pathologic examination, removing thin slices for histologic examination and segment homogenization for RNA,DNA and protein extraction.

Individual segments will be thawed on ice and homogenized immediately upon thawing. Homogenization methods will be optimized to produce the highest dissolved protein content. Methods to be trialed will include sonication, mechanical disruption by laboratory blender, mechanical disruption by manual chopping followed by Potter device, and freeze thawing.

Buffer and solvent system variables to be trialed include salt concentration, pH and buffer type, chaotrope concentration (urea and thiourea), presence of organic co-solvents such as DMSO, and the presence of nonionic detergent. All homogenization will be performed between 0 and 4°C and in the presence of protease inhibitors.

For proteomic analysis, High-performance liquid chromatography/electrospray mass spectrometry will be employed as a complementary route to discovering differences in protein expression between healthy and traumatized tissue. Following solid-phase extraction of soluble and solubilized proteins, we will optimize conditions for separation of protein peaks detected by UV absorbance and/or total ion current and may employ more than one set of conditions in order to focus on different sets of extracted proteins. We will use high-porosity C-18 reversed-phase columns to separate cytosolic proteins, and C-4 for membrane proteins. Standard methods of ionization, fragmentation, and detection will be used that are consistent with the Shimadzu LCMS-IT-TOF mass spectrometer at the Research Operations Service (ROS).

For RNA analysis, extracted RNA will be brought to the Duke Center for Genomic and Computational Biology Genomic Technologies core. There, RNA quality will be determined using an Agilent 2100bioanalyzer followed by Affymetrix GeneChip analysis. David Corcoran, the biostatistician who works at the Duke Center for Genomic and Computational Biology, will perform data analysis.

In this study, no changes to the standard of care will be implemented. The sciatic nerve specimens would otherwise be discarded as human tissue; there are no other ongoing investigations using these specimens.

Following the analysis of the sciatic nerve, we will collect data - demographic, injury, and pain treatment information, as well as pre-operative pain scores - from subjects' charts to determine secondary outcome variables. (See Appendix B - Case Report Forms)

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years and older, capable of providing informed consent indicating awareness of the investigational nature of the study, in keeping with institutional policy
* Written informed consent must be obtained from each subject prior to entering the study
* Traumatic lower extremity (above knee or below knee) amputation that occurred as a result of exposure to improvised explosive device (IED) blast, gunshot, or vehicle rollover during combat in support of OIF/OND or OEF.
* Scheduled final amputation revision to occur during the initial hospital admission at Walter Reed National Military Medical Center

Exclusion Criteria:

* Inability to provide informed consent
* Traumatic or surgical foot amputations
* Amputation occurring at Walter Reed Army Medical Center or another continental United States (CONUS) hospital after failed limb salvage
* Nerve specimen less than 5cm in length

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female Operation Iraqi Freedom (OIF)/(Operation New Dawn (OND) or Operation Enduring Freedom (OEF) veterans who meet eligibility criteria who require an amputation revision occurring during their initial hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chester c Buckenmaier, Principal Investigator — Defense and Veterans Center for Integrative Pain Management
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No